CLINICAL TRIAL: NCT06402604
Title: Stress Reduction in Formerly Preeclamptic Women; Sofa or Sports
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL78063.091.21
Record Dates: First submitted 2023-05-09; First posted 2024-05-07 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-05

CONDITIONS: Preeclampsia; Stress, Psychological; Stress, Physiological; Sports Physical Therapy
Keywords: Mindfulness Based Stress Reduction; Hair cortisol; Preeclampsia; Stress; Aerobic sports training
MeSH Terms: conditions — Pre-Eclampsia; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: One group receives a 12-weeks standard online MBSR therapy, consisting of 8 weekly group meetings, one day silent retreat, and daily homework. A second group attends a 12-week aerobe training program which consists of HR-controlled training on a cycle trainer at 70-80% individual heart rate reserve (HRR) for 2 to 3 times per week. Finally, the time control (wait list) group will be asked to continue normal activities and lifestyle and won't undergo guided mindfulness therapy or exercise training during the 12 weeks study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sports (Experimental): Exercise training consists of 12-weeks of heartrate-controlled training on a cycle trainer at 70-80% individual heartrate reserve. The training will take place at a fitness center of the participant's own choice, women will receive a sport fee after inclusion. heartrate will be monitored continuously and recorded by a smartwatch. Training is personalized and consists of 60 minutes of cycling for 2 times (week: 1-6) to 3 times (week: 7-12) per week for one hour. Training includes intensity of 40 minutes on 70-80%. heartrate reserve (HRR) was calculated in the following manner: HHR=HRmax-HRrest, in which HRmax is assumed 220 bpm minus age.
  Interventions: Behavioral: Aerobic exercise training
- Sofa (Experimental): Participants will participate in an mindfullness based stress reduction (MBSR) training. The training consists of 8 weekly sessions lasting 2,5 hours per session. A silent day of approximately 6 hours is also included, as well as daily home practice assignments of about 45 minutes. During the training participants will learn to focus their attention in the present moment in an accepting and non-judgemental way, rather than ruminating about past and future experiences. The training will be offered online and is led by qualified teachers from Radboud university medical centre.
  Interventions: Behavioral: Mindfulness Based Stress Reduction training
- Waitlist (No Intervention): The participants are asked during the intervention not to follow any diet. Women in the control group will be asked to continue normal physical activities and not to undertake Mindfulness therapy during the study period for 12 weeks.

INTERVENTIONS:
Behavioral: Aerobic exercise training — See above in arm group descriptions.
  Arms: Sports
Behavioral: Mindfulness Based Stress Reduction training — See above in arm group descriptions.
  Arms: Sofa

SUMMARY:
The goal of this clinical trial is to evaluate stress and cardiovascular risk factors in women with preeclampsia in the medical history. The main questions it aims to answer are:

* to improve our understanding of the underlying psychological and physical stress factors in relation to the circulatory risk profile in women with a history of preeclampsia
* to examine the effects of mindfullness based stress reduction (MBSR) or aerobic exercise training on hair cortisol and symptoms of mental stress.

Participants will undergo pre- and post-intervention pre-conceptional standard cardiovascular assessments, head tilt test and give a hair sample. As intervention they will sport or do mindfulness for 3 months.They will be compared with a control group.

DETAILED DESCRIPTION:
Rationale: Approximately one out of three women with pre-term preeclampsia develops a post-traumatic stress disorder or depression after pregnancy. This could be related to the psychological impact of preeclampsia and premature birth resulting in increased perceived stress. It is also possible that preeclampsia and stress levels share a common aetiology, as both appear to correlate with increased cortisol levels and higher sympathetic drive. Approximately 50% of women with a history of preeclampsia have low plasma volume levels, indicating reduced circulatory reserve. Women with a hemodynamic profile characterized by a limited circulatory reserve have increased resting sympathetic tone, and are prone to develop preeclampsia in a subsequent pregnancy. These women also report more complaints of perceived stress. This raises not only the question whether increased perceived stress in women with a history of preeclampsia originates within the brain itself (primary psychological) or whether it is a psychological reflection of underlying reduced circulatory reserves (secondary psychological), but also the question about which intervention is most effective to reduce this perceived stress level. Should the investigators focus more on the emotional coping mechanisms and psychological aspects or should the investigators aim at improving the underlying hemodynamic profile and circulatory reserves to reduce overall sympathetic drive? The investigators hypothesize that 1) both interventions in women with preeclampsia and increased mental stress complaints will result in improved circulatory reserve, lower cortisol levels, lower sympathetic resting tone, and better continuous physiological measures (as measured with a smartwatch during the trial). 2) The aerobic exercise training will additionally improve the women's cardiovascular risk profile.

Objective: To investigate the effects of online mindfulness-based stress reduction (MBSR) therapy and aerobe exercise training on mental stress, physiological stress (hair cortisol) and cardiovascular risk profile in women with a history of preeclampsia and current increased symptoms of mental stress.

Study design: Multicenter randomized trial of two interventions (online mindfulness therapy and aerobic exercise training) and a time control group who undergo neither of the two interventions (wait list group). Possible eligible women will be recruited in two tertiary hospitals (Radboudumc Nijmegen and Maastricht Medical Centre) after referral to these centres for preconceptional cardiovascular assessment after severe preeclampsia in a previous pregnancy. Participants with symptoms of mental stress will be randomly assigned to either one of the two intervention groups or the wait list (3 options) after the Preconceptional Cardiovascular Assessment (PcCA) and Stress Assessment (SA). After 12 weeks of intervention, or in the case of the wait list group, 12 weeks without intervention, another PcCA and SA will take place. Results after 12 weeks will be compared with baseline results. Additionally, in all groups online questionnaires will be filled in 6 months after baseline assessments. Women who were allocated to the wait list group are offered either mindfulness therapy or aerobic exercise training after completing the second PcCA and SA after 12 weeks.

Study population: Primiparous women with an obstetric history of preeclampsia, according to ISSHP definition, who score ≥ 16 on the Perceived Stress Scale (PSS) ≥ 41 on the State-Trait Anxiety Inventory (STAI) or ≥ 10 on the Edinburgh Postnatal Depression Scale (EPDS) during online questionnaires as part of the anamnesis of PcCA will be prompted to join the study. Women with pre-existent diabetes mellitus, autoimmune disease, overt cardiovascular disease, or use of tabacco or medication that might affect the cardiovascular system are excluded from participation. Other exclusion criteria are plans to become pregnant within the time frame of the intervention (12 weeks) at time of baseline assessment.

Intervention: One group receives a 12-weeks standard online MBSR therapy, consisting of 8 weekly group meetings, one day silent retreat, and daily homework. A second group attends a 12-week aerobe training program which consists of HR-controlled training on a cycle trainer at 70-80% individual heart rate reserve (HRR) for 2 to 3 times per week. Finally, the time control (wait list) group will be asked to continue normal activities and lifestyle and won't undergo guided mindfulness therapy or exercise training during the 12 weeks study period.

Main study parameters: The primary endpoint is mental stress, evaluated with validated questionnaires PSS, STAI and EPDS. Secondary endpoints are the results of pre- and post-intervention pre-conceptional standard cardiovascular assessments. These cardiovascular assessments are in Maastricht UMC+ tertiary hospital care as usual after referral for preconceptional evaluation in women with a history of preeclampsia. This assessment includes: biometrics, 30-minutes blood pressure and heart rate measurement, venous blood samples for metabolic syndrome screening, echocardiography and plasma volume assessment. For this specific study the investigators will additionally assess cortisol concentration in hair and evaluate sympathetic activity during a head-up tilt test using non-invasive heart rate variability analysis. During the exercise training, heartbeat monitoring will be measured using smartwatches. Feasibility of the interventions will be evaluate with additional participant survey at follow-up measurement.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given
* Age > or = 18 years
* Good understanding of Dutch language
* Preeclampsia in prior pregnancy, defined as the combination of gestational hypertension (≥140/90 mmHg, measured twice, six hours or more apart), and proteinuria (consistently ≥300mg/24 hours) after 20 weeks of pregnancy in previously normotensive women, according to International Society for the Study of Hypertension in Pregnancy (Brown, 2018).
* Normotensive at the time of baseline measurements
* Perceived Stress Scale score ≥ 16 or State-Trait Anxiety Inventory (STAI) score ≥ 41 or Edinburgh Postnatal Depression Scale (EPDS) score ≥ 10

Exclusion Criteria:

* Pre-existent diabetes mellitus, autoimmune disease, HIV positivity or overt cardio-vascular disease.
* Use of medication or supplements that might affect the cardiovascular system
* (Physical) inabilities to complete 12 weeks of moderate exercise training
* Currently involved in psychological therapy or mindfullness training.
* Pregnancy
* Women who intend to become pregnant within 12 weeks after baseline assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women with obstetric history.
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Perceived stress | Pre-post intervention and 3 months follow up.
  according to the measures on Perceived Stress Scale,minimum 0, maximum 40. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Anxiety symptoms | Pre-post intervention and 3 months follow up.
  according to the measures on State-Trait Anxiety Inventory, Scores range from 20 to 80, with higher scores correlating with greater anxiety. Score above 40 represents significant anxiety symptoms
Depression symptoms | Pre-post intervention and 3 months follow up.
  according to the measures on postnatal Depression Scale. Scores range from 0 to 30, with higher scores correlating with more depression symptoms. Score above 10 represents significant depression.

SECONDARY OUTCOMES:
Weight | Pre-post intervention of 3 months.
  weight in kilograms
Height | Pre-post intervention of 3 months.
  height in meters
body surface area | Pre-post intervention of 3 months.
  body surface area (BSA) was calculated using the Dubois & Dubois formula
30-minutes blood pressure and heart rate measures | Pre-post intervention of 3 months.
  systolic and diastolic pressure in mmHg, heart reat in beat/min
Sympathetic activity | Pre-post intervention of 3 months.
  Sympathetic activity was measured using the head-up tilt test (HUT) using a finometer. During this test orthostatic stress was tested to assess the changes in sympathetic activity.
glucose | Pre-post intervention of 3 months.
  in mmol/L, venous blood samples for metabolic parameters were drawn in fasting state
insulin | Pre-post intervention of 3 months.
  in mU/l, venous blood samples for metabolic parameters were drawn in fasting state
total cholesterol | Pre-post intervention of 3 months.
  Venous blood samples for metabolic parameters were drawn in fasting state
lowdensity lipoprotein cholesterol | Pre-post intervention of 3 months.
  Venous blood samples for metabolic parameters were drawn in fasting state
high-density lipoprotein cholesterol | Pre-post intervention of 3 months.
  Venous blood samples for metabolic parameters were drawn in fasting state
triglycerides | Pre-post intervention of 3 months.
  in mmol/L, venous blood samples for metabolic parameters were drawn in fasting state
renal function | Pre-post intervention of 3 months.
  Venous blood sample for serum creatinine levels (in μmol/L).
Urine sample | Pre-post intervention of 3 months.
  protein per liter
Plasma volume | Pre-post intervention of 3 months.
  in ml, was measured by using the 125I-Human Serum Albumin indicator dilution technique (125I-has). It was calculated by dividing the total injected 125I-has by the virtual volume-specific radioactivity at time zero (31). Eventually plasma volume was calculated by dividing total plasma volume by BSA, resulting in ml/m2 (24).
Hair cortisol concentration | Pre-post intervention of 3 months.
  cortisol in hair.

OTHER OUTCOMES:
Age | Pre-intervention.
  in years
highest education | Pre-intervention.
  highest education
Smoking | Pre-intervention.
  tabaco use
Smoking | Pre-intervention.
  tabacco use
Alcohol | Pre-intervention.
  alcohol use
Drugs | Pre-intervention.
  drug use
Obstetric history | Pre-intervention.
  description of previous pregnancy outcome
Patient hair properties | Pre-intervention.
  Hair properties: color, treatments and wash frequency
Comorbidities | Pre-intervention.
  medical history
use of medication | Pre-intervention.
  medication use
Physical activity evaluation | Pre-post intervention and 3 months follow up.
  Short Questionaire to assess health enhancing physical activity (SQUASH), to asses physical activity in a week including, actively commuting (walking, cycling), physical activity at work or school, household activities, leisure time activities (sports, walking, gardening, cycling). The higher the score, the higher the more time is spend to physical activity.
Mindfulness and self-awareness | Pre-post intervention and 3 months follow up.
  (The Five Facet Mindfulness Questionnaire, FFMQ-SF) minimum 15 and maximum score.75. The higher the score, the more attention for participant to be here and now.
Heart rate | Pre-post intervention of 3 months.
  Heart rate during aerobe exercise training, divided in HR-zones

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Joris J.A. van Esch, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data available on request.